CLINICAL TRIAL: NCT05816343
Title: Long Term Efficacy and Safety of Orlistat for Type 1 Hyperlipoproteinemia: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Long Term Efficacy and Safety of Orlistat for Type 1 Hyperlipoproteinemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Abhimanyu Garg, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: STU-2019-0776
Record Dates: First submitted 2023-04-01; First posted 2023-04-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Hyperlipoprotenemia
MeSH Terms: interventions — Orlistat

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, parallel, study design will be employed for the first 24 weeks (Phase 1) followed by an open-labeled period of 24 weeks (Phase 2).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orlistat Drug (Active Comparator): Drug will be given orally.
  Interventions: Drug: Orlistat
- Placebo (Placebo Comparator): Placebo will be given orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orlistat — Orlistat is an inhibitor of gastric and pancreatic lipases and can reduce dietary fat absorption by 30%. Orlistat at a dose of 2 capsules (each containing 60 mg of active drug) three times a day with each meal (a total dose of 360 mg daily).
  Other Names: Alli
  Arms: Orlistat Drug
Drug: Placebo — Placebo at a dose of 2 capsules (each containing 60 mg placebo) three times a day with each meal (a total dose of 360 mg daily).
  Arms: Placebo

SUMMARY:
Type I hyperlipoproteinemia (T1HLP, also known as familial chylomicronemia syndrome or FCS) is a rare diseasewhere the blood triglycerides (fats) are very high. It is caused by lack of certain enzymes and proteins in the bodythat are important in disposing circulating fats from blood. Treatment of T1HLP patients who have very high levels of blood fats (≥ 1,000 mg/dL) is challenging as conventional triglyceride-lowering medications, such as fibrates and fishoil, are ineffective.

The purpose of this trial is to study the long-term efficacy and safety of orlistat for reducing blood triglyceride levels in patients with T1HLP.

DETAILED DESCRIPTION:
The hypotheses to be tested and the specific aims are:

Hypothesis 1: As compared to placebo, Orlistat will be effective and safe in lowering fasting serum TG concentrations in patients with T1HLP.

Specific Aim 1: To investigate the efficacy and safety of Orlistat for reducing fasting serum TG levels in 28 patients with T1HLP in a double-blind, randomized, placebo-controlled, parallel design study for a period of 24 weeks.

Hypothesis 2: The efficacy and safety of Orlistat in patients with T1HLP will be maintained over a period of up to 48 weeks.

Specific Aim 2: To investigate the efficacy and safety of Orlistat in patients with T1HLP in an open-label extension study for a period of up to 48 weeks-.

After a screening evaluation, the subjects will be advised to consume an extremely low fat diet (≤15% of total energy from fat) for the entire duration of the study. After the baseline period of 8 weeks, they will be randomly assigned to placebo or Orlistat for the duration of 24 weeks (Phase 1). After Phase 1, all patients will enter an open-label extension (Phase 2) and receive Orlistat for a period of 24 weeks for a total study duration of 56 weeks. During the last week of Baseline Period, Phase 1, and Phase 2, blood lipids and chemistry panel will be analyzed for three consecutive days, and fat-soluble vitamin levels will be measured once. All the visits are going to be outpatient.

ELIGIBILITY:
* Type I hyperlipoproteinemia confirmed by bi-allelic disease-causing variants in any one of the T1HLP genes (LPL, APOC2, APOA5, LMF1, GPIHBP1, or GCKR).
* Subjects who have a fasting TG greater than or equal to 750 mg/dL at the end of run-in period of 8 weeks will be eligible for randomization.
* Age ≥ 8 years
* Well controlled diabetes mellitus with hemoglobin A1c < 8%
* Off orlistat for a period of 2 months

Exclusion Criteria:

* Secondary hypertriglyceridemia due to diabetes, renal disease, , alcoholism and drug therapy such as estrogens and estrogen analogues, steroids, HIV-1 protease inhibitors, retinoic acid derivatives, interferons, or lasparaginase.
* On lomitapide or participating in clinical trial of volanesorsen and olezarsen
* On cyclosporine
* Having serum TSH outside of the normal range if on levothyroxine supplementation.
* Use of levothyroxine to suppress TSH in individuals with thyroid cancer.
* Pregnant or lactating women
* Significant liver disease (elevated transaminases > 2 times upper limit of normal)
* Alcohol abuse (> 7 drinks or 84 g per week for women and > 14 drinks or 168 g per week for men)
* Severe anemia (hematocrit < 24%)
* Illicit drug use (cocaine, marijuana, LSD, etc.)
* Major surgery in the past three months
* Congestive heart failure
* Serum creatinine greater than 2.5 mg/dL
* Cancer within the past five years
* Gastrointestinal surgery in the past
* Current therapy with anti-coagulants, digoxin and anti-arrhythmics
* Chronic malabsorption syndromes
* Cholestasis
* Acute illnesses such as acute pancreatitis in the last 8 weeks
* Previous history of renal calcium oxalate stones

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Triglycerides | 24 weeks
  Change in fasting serum TG levels weeks compared to the baseline fasting serum TG levels .

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu G Garg, MD, Principal Investigator — University of Texas Southwestern Medical Center; Chandna Vasandani, Ph.D, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- UT southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided